CLINICAL TRIAL: NCT07315906
Title: Investigation of the Acute Effects of Different Physiotherapy Methods Applied to the Patellar Tendon: A Single-Blind Randomized Controlled Trial
Brief Title: Patellar Tendon Physiotheraphy Acute Effects Trial
Acronym: PTPAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Elif Akduran, Principal İnvestigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTT-2025-DEU
Record Dates: First submitted 2025-12-21; First posted 2026-01-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Patellar Tendon
Keywords: patellar tendon; physiotheraphy; deep friction massage; thermal imaging; quadriceps exercise; muscle strength; thermography; flexibility; tendon temperature; healthy adults; tendon physiology; acute effects; knee biomechanics; patellar tendinitis; Patellar tendon pain; physical therapy modalities

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of four parallel groups, each receiving a single physiotherapy intervention or no intervention. The study used a randomized parallel design to compare acute responses among the four groups.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Deep Friction Massage (Experimental): A single session of deep friction massage applied directly to the patellar tendon
  Interventions: Other: Deep Friction Massage
- Thermal Agent Application (Experimental): A locally applied superficial thermal agent delivered as a single session.
  Interventions: Other: Thermal Agent Application
- Quadriceps Exercise (Experimental): A single session of standardized quadriceps resistance exercise protocol.
  Interventions: Other: Quadriceps Exercise
- Control (No Intervention): No treatment administered; participants remained at rest during the session.

INTERVENTIONS:
Other: Deep Friction Massage — A single session of deep friction massage applied directly to the patellar tendon.
  Arms: Deep Friction Massage
Other: Thermal Agent Application — A single application of a thermal agent (hot pack) applied to the patellar tendon region.
  Arms: Thermal Agent Application
Other: Quadriceps Exercise — A single session of quadriceps resistance exercise targeting knee extensor muscles.
  Arms: Quadriceps Exercise

SUMMARY:
This randomized controlled trial investigated the acute effects of different physiotherapy interventions applied to the patellar tendon. Participants were randomly assigned to one of four groups: deep friction massage, thermal agent application, quadriceps resistance exercise, or a control group. Each intervention was delivered in a single session. Outcomes of the study included changes in skin temperature, muscle strength, flexibility, and pulse rate. All measurements were taken immediately before the intervention and again immediately after, 15 minutes after, and 60 minutes after the intervention. The study was conducted with healthy adult volunteers. The results of this study are expected to contribute to a better understanding of how different physiotherapy modalities acutely influence the patellar tendon region.

DETAILED DESCRIPTION:
This study examined the immediate physiological responses of the patellar tendon region following different physiotherapy interventions. Participants were allocated into four groups: (1) deep friction massage applied directly to the patellar tendon, (2) a locally applied superficial thermal agent, (3) a structured quadriceps resistance exercise protocol, and (4) a no-intervention control group. Each intervention was administered as a single session under standardized laboratory conditions.

Outcome measures included skin temperature assessed with thermal imaging, quadriceps muscle strength measured with a handheld dynamometer, flexibility assessed by standardized clinical procedures, and pulse rate. All measurements were collected at four time points: immediately before the intervention, immediately after, 15 minutes after, and 60 minutes after the intervention.

The study was conducted with healthy adult volunteers to evaluate the acute physiological effects of commonly used physiotherapy modalities on the patellar tendon region. The findings are intended to inform clinical decision-making by clarifying how different physiotherapy techniques influence tendon-related parameters within the first hour following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 24 years
* Not having engaged in regular exercise training within the past 6 months
* Body Mass Index (BMI) below 30
* Ability to complete all assessment procedures
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Presence of any systemic or musculoskeletal disorder
* Onset of pain during the assessment procedure
* History of knee joint or peri-articular injury within the past 6 months
* Presence of neurological, vascular, or rheumatological disease
* Any dermatological condition that may affect skin integrity

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Skin Temperature Change | Baseline, immediately after intervention, 15 minutes after, 60 minutes after
  Skin temperature of the patellar tendon region measured using infrared thermography at four time points to analyze acute thermal response.
Quadirceps Muscle Strength | Baseline, immediately after intervention, 15 minutes after, 60 minutes after
  Isometric quadriceps muscle strength measured with a handheld dynamometer at four time points to assess acute changes following intervention.
Hamstring and Quadriceps Flexibility | Baseline, immediately after intervention, 15 minutes after, 60 minutes after
  Flexibility of the quadriceps and hamstring assessed using a standardized stretching test at four time points to assess evaluate changes.
Dorsalis Pedis Pulse Rate | Baseline, immediately after intervention, 15 minutes after, 60 minutes after
  Pulse rate measured by palpation at four time points (baseline, immediately after intervention, 15 minutes, and 60 minutes) to evaluate acute cardiovascular response to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, İzmir, Izmir, balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No